CLINICAL TRIAL: NCT01706796
Title: A Phase 1, Open Label, Randomized, Single Dose, 5 Period Crossover Relative Bioavailability Study In Healthy Volunteers Evaluating Spray Dried Dispersion (SDD) Immediate Release (IR) PF-06273340 Tablet, Two SDD Modified Release (MR) Matrix Tablets In Comparison With PF-06273340 Oral Solution, Including Preliminary Assessment Of Food Effect
Brief Title: A Study Comparing PF-06273340 Immediate Release Tablet, PF-06273340 Modified Release Tablets To PF-06273340 Oral Solution In The Fasted State. This Study Will Also Compare PF-06273340 Modified Release Tablets In Fasted And Fed State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B5261003
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Pain
MeSH Terms: conditions — Pain | interventions — PF-06273340

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- PF-06273340 Oral Solution Fasted (Experimental)
  Interventions: Drug: PF-06273340
- PF-06273340 Immediate Release Tablet Fasted (Experimental)
  Interventions: Drug: PF-06273340
- PF-06273340 Modified Release (MR1) Tablet Fasted (Experimental)
  Interventions: Drug: PF-06273340
- PF-06273340 Modified Release (MR2) Tablet Fasted (Experimental)
  Interventions: Drug: PF-06273340
- PF-06273340 Modified Release (MR1) Tablet Fed (Experimental)
  Interventions: Drug: PF-06273340
- PF-06273340 Modified Release (MR2) Tablet Fed (Experimental)
  Interventions: Drug: PF-06273340

INTERVENTIONS:
Drug: PF-06273340 — Oral solution, single dose, fasted
  Arms: PF-06273340 Oral Solution Fasted
Drug: PF-06273340 — Immediate Release Tablet, single dose, fasted
  Arms: PF-06273340 Immediate Release Tablet Fasted
Drug: PF-06273340 — Modified Release Tablet (short duration, MR1), single dose, fasted
  Arms: PF-06273340 Modified Release (MR1) Tablet Fasted
Drug: PF-06273340 — Modified Release Tablet (long duration, MR2), single dose, fasted
  Arms: PF-06273340 Modified Release (MR2) Tablet Fasted
Drug: PF-06273340 — Modified Release Tablet (short duration, MR1), single dose, fed
  Arms: PF-06273340 Modified Release (MR1) Tablet Fed
Drug: PF-06273340 — Modified Release Tablet (long duration, MR2), single dose, fed
  Arms: PF-06273340 Modified Release (MR2) Tablet Fed

SUMMARY:
The primary purpose of this study is to estimate the relative bioavailability and food effect of PF-06273340 tablets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-child bearing potential, between the ages of 21 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* Screening supine blood pressure >=140 mm Hg (systolic) or >=90 mm Hg (diastolic), on a single measurement (confirmed by a single repeat, if necessary) following at least 5 minutes of rest.
* Evidence or history of orthostatic hypotension.
* 12-lead ECG demonstrating QTc >450 or a QRS interval >120 msec at Screening. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility.
* Pregnant or nursing females; females of childbearing potential, including those with tubal ligation.
* Use of prescription or nonprescription drugs, vitamins and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Herbal supplements must be discontinued 28 days prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of <=1 g/day. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Unwilling or unable to comply with the Lifestyle guidelines described in this protocol.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Subjects who are investigational site staff members or relatives of those site staff members or subjects who are Pfizer employees directly involved in the conduct of the trial.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | up to 48 h post dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | up to 48 h post dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | up to 48 h post dose
Elimination half life | up to 48 h post dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | up to 48 h post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5261003&StudyName=A%20Study%20Comparing%20PF-06273340%20Immediate%20Release%20Tablet%2C%20PF-06273340%20Modified%20Release%20Tablets%20To%20PF-06273340%20Oral%20Solution%20In%20The%20Fasted%20